CLINICAL TRIAL: NCT01947686
Title: Survivorship and Outcomes of Robotically Assisted Patellofemoral UKA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: St. Helena Hospital Coon Joint Replacement Institute (Other)
Collaborators: Rebound Orthopedics and Neurosurgery (Unknown)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Patellofemoral Knee Arthroplasty
Keywords: osteoarthritis, patellofemoral
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patellofemoral Knee Arthroplasty: Patient who have received a robotically guided isolated patellofemoral implant.
  Interventions: Device: Robotically guided patellofemoral UKA isolated patellofemoral implants

INTERVENTIONS:
Device: Robotically guided patellofemoral UKA isolated patellofemoral implants — A robot guided isolated patellofemoral unicompartmental knee arthroplasty procedures to replace only the patellofemoral component of the knee.

SUMMARY:
The purpose of the study is to determine the survivorship rate of robotically guided isolated patellofemoral implants at 2, 5 and 10 year postoperative.

DETAILED DESCRIPTION:
The purpose of the study is to determine the survivorship rate of robotically guided isolated patellofemoral implants at 2, 5 and 10 year postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Over 21 years of age underwent primary robotically guided UKA and received an isolated patellofemoral implant at least 24 months post operative as of February 2013

Exclusion Criteria:

* Patient will be excluded from participation in the study if they are cognitively unable to answer study questions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a primary robotically guided UKA and received an isolated patellofemoral implant.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
10 year survivorship of robotically guided isolated patellofemoral implants. | 10 years after surgery
  10 year survivorship of robotically guided isolated patellofemoral implants at 2,5, and 10 year follow up.

SECONDARY OUTCOMES:
2 year survivorship of robotically guided isolated patellofemoral implants. | 2 years after surgery
  The survivorship rate of robotically guided isolated patellofemoral implants at 2,5, and 10 year.
5 year survivorship of robotically guided isolated patellofemoral implants. | 5 years after surgery
  The survivorship rate of robotically guided isolated patellofemoral implants at 2,5, and 10 years post operative.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Coon, MD, Study Director — St. Helena Hospital Coon Joint Replacement; Todd Borus, MD, Principal Investigator — Rebound Orthopedics and Neurosurgery
Locations (2):
- United States (2):
  - St. Helena Hospital Coon Joint Replacement Institute, St. Helena, California
  - Rebound Orthopedics and Neurosurgery, Vancouver, Washington